CLINICAL TRIAL: NCT02192515
Title: A Phase 1 Study of APD356 (Lorcaserin) in Healthy Japanese Adult Subjects
Brief Title: A Study of APD356 (Lorcaserin) in Healthy Japanese Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APD356-J081-101
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Healthy Subjects
Keywords: Healthy Subjects; Japanese Adult
MeSH Terms: interventions — lorcaserin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- APD356 10 mg (Experimental): Subjects will be randomized to APD356 10 mg group (6 subjects) or placebo group (2 subjects) to receive single dose of study drug.
  Interventions: Drug: APD356 10 mg; Drug: APD356 10 mg matching Placebo
- APD356 20 mg (Experimental): Subjects will be randomized to APD356 20 mg group (6 subjects) or placebo group (2 subjects) to receive single dose of study drug.
  Interventions: Drug: APD356 20 mg; Drug: APD356 20 mg matching Placebo
- APD356 XR-20 mg (Experimental): Subjects will be randomized to APD356 XR-20 mg group (6 subjects) or placebo group (2 subjects) to receive single dose of study drug on Day 1 and multiple doses of study drug on Day 8-14 once daily before breakfast.
  Interventions: Drug: APD356 XR-20 mg; Drug: APD356 XR-20 mg matching Placebo
- APD356 10 mg and APD356 XR-20mg (orange tablet) (Experimental): Subjects will be randomized to Sequence A (8 subjects) or Sequence B (8 subjects) to receive study drug in the sequence shown below.
  Sequence A: 10 mg tablet, 2 doses (12 hours apart) => XR-20 mg orange tablet, single dose => XR-20 mg orange tablet, q. d., multiple doses (fasted) => XR-20 mg orange tablet, q. d., multiple dose (fed)
  Sequence B: XR-20 mg orange tablet, single dose => 10 mg tablet, 2 doses (12 hours apart) => XR-20 mg orange tablet, q. d., multiple dose (fed) => XR-20 mg orange tablet, q. d., multiple doses (fasted)
  Interventions: Drug: APD356 10 mg; Drug: APD356 XR-20 mg (orange tablet); Drug: APD356 XR-20mg (orange tablet, fed state)

INTERVENTIONS:
Drug: APD356 10 mg — One tablet of APD356 10 mg will be orally administered in fasted state.
  Arms: APD356 10 mg; APD356 10 mg and APD356 XR-20mg (orange tablet)
Drug: APD356 XR-20 mg — One tablet of APD356 XR-20 mg will be orally administered in fasted state.
  Arms: APD356 XR-20 mg
Drug: APD356 10 mg matching Placebo — One tablet of APD356 10 mg matching placebo will be orally administered in fasted state.
  Arms: APD356 10 mg
Drug: APD356 XR-20 mg matching Placebo — One tablet of APD356 XR matching placebo will be orally administered in fasted state.
  Arms: APD356 XR-20 mg
Drug: APD356 20 mg — Two tablets of APD356 10 mg will be orally administered in fasted state.
  Arms: APD356 20 mg
Drug: APD356 20 mg matching Placebo — Two tablets of APD356 10 mg matching placebo will be orally administered in fasted state.
  Arms: APD356 20 mg
Drug: APD356 XR-20 mg (orange tablet) — One tablet of APD356 XR-20 mg orange tablet will be orally administered in fasted state.
  Arms: APD356 10 mg and APD356 XR-20mg (orange tablet)
Drug: APD356 XR-20mg (orange tablet, fed state) — One tablet of APD356 XR-20 mg orange tablet will be orally administered 30 minutes after the start of a meal.
  Arms: APD356 10 mg and APD356 XR-20mg (orange tablet)

SUMMARY:
The purpose of this study is to assess the safety and pharmacokinetics of APD356 in healthy Japanese adult subjects. Regarding cohorts 1 to 3, this study is a single center, placebo-controlled, randomized,double-blind study. Regarding cohort 4, this study is a single center, randomized, open-label study that consists of two sequential two-way crossover studies. The study consists of 4 cohorts. In cohort 1, subjects will be randomized to 10 mg group (6 subjects) or placebo group (2 subjects) to receive single dose of study drug. In cohort 2, subjects will be randomized to 20 mg group (6 subjects) or placebo group (2 subjects) to receive single dose of study drug. In cohort 3, subjects will be randomized to XR-20 mg group (6 subjects) or placebo group (2 subjects) to receive single dose of study drug on Day 1 and multiple doses of study drug on Day 8-14 once daily before breakfast. In cohort 4, subjects will be randomized to Sequence A (8 subjects) or Sequence B (8 subjects) to receive study drug in the sequence shown below.

Sequence A: 10 mg tablet, 2 doses (12 hours apart) => XR-20 mg orange tablet, single dose => XR-20 mg orange tablet, q. d., multiple doses (fasted) => XR-20 mg orange tablet, q. d., multiple dose (fed)

Sequence B: XR-20 mg orange tablet, single dose => 10 mg tablet, 2 doses (12 hours apart) => XR-20 mg orange tablet, q. d., multiple dose (fed) => XR-20 mg orange tablet, q. d., multiple doses (fasted)

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all of the following criteria to be included in this study:

1. Non-smoking, healthy Japanese male subjects age greater than or equal to 20 years and less than 55 years old at the time of informed consent. To be considered non-smokers, subject must have discontinued smoking for at least 4 weeks prior to dosing.
2. BMI greater than or equal to 23 and less than 32 kg/m2 at Screening

   a) BMI (kg/m2) = body weight(kg)/[height(m) x height(m)]
3. Provide written informed consent
4. Willing and able to comply with all aspects of the protocol

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

1. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing
2. Evidence of disease that may influence the outcome of the study within 4 weeks prior to dosing; eg, psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or subjects who have a congenital abnormality in metabolism
3. Any history of gastrointestinal surgery that may affect PK profiles of study drug, eg, hepatectomy, nephrotomy, digestive organ resection at Screening
4. Any clinically abnormal symptom or organ impairment found by medical history at Screening, and physical examinations, vital signs, ECG finding, or laboratory test results that require medical treatment at Screening
5. A prolonged QT/QTc interval (QTc greater than 450 ms) demonstrated on ECG at Screening or Baseline
6. Known history of clinically significant drug allergy at Screening
7. Known history of food allergies or presently experiencing significant seasonal or perennial allergy at Screening
8. Known to be human immunodeficiency virus (HIV) positive at Screening
9. Positive results for Hepatitis B surface antigen (HBs Ag), Hepatitis C virus antibody (HCV Ab) or Syphilis test at Screening
10. History of drug or alcohol dependency or abuse, or those who have a positive urine drug test at Screening or Baseline
11. Intake of caffeinated beverages or food within 72 hours prior to dosing
12. Intake of nutritional supplements, juice, and herbal preparations or other foods or beverages that may affect the various drug metabolizing enzymes and transporters (eg, alcohol and grapefruit juice) within 1 week prior to dosing
13. Intake of herbal preparations containing St. John's Wort within 4 weeks prior to dosing
14. Use of prescription drugs (except for disinfectants, eye drops) within 4 weeks prior to dosing
15. Intake of over-the-counter (OTC) medications (except for disinfectants, eye drops) within 2 weeks prior to dosing
16. Currently enrolled in another clinical study or used any investigational drug or device within 16 weeks preceding informed consent
17. Subjects who undergo blood transfusion within 12 weeks, or who donate 400 mL or more of whole blood within 12 weeks (16 weeks for woman) or 200 mL or more of whole blood within 4 weeks, or who make a component donation within 2 weeks prior to dosing.
18. Engagement in strenuous exercise within 2 weeks prior to check-in (eg, marathon runners, weight lifters, etc.)
19. Subjects who have any condition that would make them, in the opinion of the investigator, unsuitable for the study

Ages: 20 Years to 54 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-07; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by adverse events (AEs), clinical laboratory tests, vital signs, body weight and ECGs | Up to 30 days after last dose
Pharmacokinetics of APD356: Cmax | Up to 96 hours after last dose
Pharmacokinetics of APD356: tmax | Up to 96 hours after last dose
Pharmacokinetics of APD356: AUC | Up to 96 hours after last dose
Pharmacokinetics of APD356: t1/2 | Up to 96 hours after last dose

CONTACTS AND LOCATIONS:
Locations (1):
- Toshima-Ku, Tokyo, Japan